CLINICAL TRIAL: NCT03480386
Title: Home Pulmonary Rehabilitation for COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Roberto P. Benzo, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-009449; R01HL140486-01 (NIH)
Record Dates: First submitted 2018-02-26; First posted 2018-03-29 (Actual); Results first posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Emphysema
Keywords: Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Intervention Model Description: Randomization will be stratified by whether the participant has poor lung function (forced expiratory volume [FEV1] <50% predicted) and whether the participant has severe dyspnea (recorded modified Medical Research Council Dyspnea Scale [mMRC] score, 3-4; scale, 0-4); critical factors that can make the study arms unbalanced regarding risk factors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Rehabilitation Program Intervention (Experimental): Subjects will receive 12 weeks home pulmonary rehabilitation (PR) with health coaching.
  Interventions: Behavioral: Home Based Pulmonary Rehabilitation
- Usual Care (No Intervention): Subjects will receive 12 weeks of usual care.

INTERVENTIONS:
Behavioral: Home Based Pulmonary Rehabilitation — Twice daily exercise routine six days a week of 3 minutes of personal breathing, 5 exercises with 10 reps each, and 6 minutes of walking with weekly health coach calls.
  Arms: Pulmonary Rehabilitation Program Intervention

SUMMARY:
Regular physical activity has been found to be important in maintaining health and well-being in people with COPD. The purpose of this study is to test new technology and health coaching aimed to help people with COPD become more physically active in their daily lives.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD, confirmed by spirometry
* Age ≥40 years (to avoid recruiting participants with asthma rather than COPD)
* Current or previous smoker (≥10 packs per year)
* Confidence in using the proposed pulmonary rehabilitation (PR) system
* English language fluency

Exclusion Criteria:

* Study candidate experiencing an acute COPD exacerbation (can be included after the acute event)
* Inability to walk (orthopedic-neurologic problems or confined to a bed)
* Currently in PR or finished PR in the last three months (unlikely to improve)
* Pregnant women
* Live in an area where cell phones do not work/

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto P Benzo, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Health Partners, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Result] Benzo R, Hoult J, McEvoy C, Clark M, Benzo M, Johnson M, Novotny P. Promoting Chronic Obstructive Pulmonary Disease Wellness through Remote Monitoring and Health Coaching: A Clinical Trial. Ann Am Thorac Soc. 2022 Nov;19(11):1808-1817. doi: 10.1513/AnnalsATS.202203-214OC. PMID 35914215
- [Derived] Benzo M, Lee M, Clark MM, Benzo R. The Basic Science of Behavior Change in COPD: Testing Self-Determination Theory to Support Home-Based Rehabilitation With Health Coaching. J Cardiopulm Rehabil Prev. 2025 Jul 1;45(4):286-293. doi: 10.1097/HCR.0000000000000957. Epub 2025 Jun 26. PMID 40476761
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pulmonary Rehabilitation Program Intervention | Usual Care
Started | 188 | 187
Completed | 143 | 142
Not Completed | 45 | 45
Not completed — Did not complete measures at 3-months | 17 | 14
Not completed — No baseline measures | 11 | 14
Not completed — Death | 0 | 5
Not completed — Withdrawal by Subject | 12 | 8
Not completed — Lost to Follow-up | 2 | 1
Not completed — Complicating disease | 0 | 1
Not completed — Disease progression | 3 | 0
Not completed — Became ineligible | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulmonary Rehabilitation Program Intervention | Usual Care | Total
Number analyzed (Participants) | 188 | 187 | 375
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.335 (9.530) | 68.676 (9.530) | 69 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 111 | 212
  Male | 87 | 76 | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 181 | 181 | 362
  Unknown or Not Reported | 5 | 5 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 177 | 180 | 357
  Black or African American | 3 | 5 | 8
  Asian | 2 | 0 | 2
  American Indian/Alaska Native | 2 | 0 | 2
  Native Hawaiian/Other Pacific Islander | 1 | 0 | 1
  More than One Race | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 188 | 187 | 375

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life
Description: The Chronic Respiratory Questionnaire (CRQ) is a validated tool, completed by participants at baseline and 3 months and measured health-related quality of life. This questionnaire measures both physical and emotional aspects of chronic respiratory disease. All scores have a range of 1 to 7, a higher number being better health-related quality of life. We reported the difference between baseline and 3 months on the CRQ emotional summary score (comprised of the mastery and emotional domains) and the physical summary score (comprised of dyspnea and fatigue domains). 0.5 points is the minimal clinically important difference for this tool.
Time Frame: Baseline, 3 months
Population: Intent-to-treat analyses, if a month three measure is missing for any reason, it will be described as not changing from baseline.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pulmonary Rehabilitation Program Intervention | Usual Care
Number analyzed (Participants) | 142 | 142
score on a scale
  CRQ Physical | 0.37 [0.24 to 0.51] | -0.17 [-0.29 to 0.05]
  CRQ Emotional | 0.43 [0.29 to 0.57] | -0.08 [-0.2 to 0.05]

2. Secondary Outcome: Change in Self-management Abilities
Description: Measured using the Self-Management Ability Scale-30 item questionnaire to assess ability and function. The SMAS consists of 30 items on four- and five-point Likert scales. Total score ranging from 0 to 100 with higher score indicating a higher function and ability, better outcome.
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pulmonary Rehabilitation Program Intervention | Usual Care
Number analyzed (Participants) | 144 | 142
score on a scale | 3.84 [2.44 to 5.24] | 0.54 [-0.62 to 1.71]

3. Secondary Outcome: Change in Physical Activity
Description: The change in average daily activity (measured in minutes) for the top 3 to 5 most active days during the measured period. Measured by the Actigraph GT3X .
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Pulmonary Rehabilitation Program Intervention | Usual Care
Number analyzed (Participants) | 128 | 138
minutes
  Daily Light Physical Activity | 17.51 [4.54 to 30.49] | 0.6 [-13.22 to 14.42]
  Daily Moderate Physical Activity | 4.47 [-3.17 to 12.11] | -4.82 [-11.66 to 2.01]
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program Intervention vs Usual Care; Daily Light Physical Activity; Test type: Superiority; p = 0.0788, t-test, 2 sided
Statistical Analysis 2: Comparison: Pulmonary Rehabilitation Program Intervention vs Usual Care; Daily Moderate Physical Activity; Test type: Superiority; p = 0.0742, t-test, 2 sided

4. Secondary Outcome: Change in Daily Step Counts
Description: Measured by the Actigraph wGT3X-BT worn for 7 days continuously to measure daily step count.
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: steps/day
Arm/Group | Pulmonary Rehabilitation Program Intervention | Usual Care
Number analyzed (Participants) | 128 | 138
steps/day | 478.63 [108.02 to 849.25] | -146.53 [-458.5 to 165.44]
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program Intervention vs Usual Care; Test type: Superiority; p = 0.0113, t-test, 2 sided

5. Secondary Outcome: Change in Depression
Description: Measured by the Patient Health Questionnaire-9 item questionnaire screening for depression. Total score range from 0 to 27. A higher score indicates that depression may be present.
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pulmonary Rehabilitation Program Intervention | Usual Care
Number analyzed (Participants) | 144 | 142
score on a scale | -1.12 [-1.67 to -0.58] | 0.08 [-0.46 to 0.62]
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program Intervention vs Usual Care; Test type: Superiority; p = 0.0021, t-test, 2 sided

6. Secondary Outcome: Social Support
Description: Measured by the Interpersonal Support Evaluation List (ISEL-12) a 12-item measure of perceptions of social support utilizing three different subscales designed to measure three dimensions of f perceived social support (appraisal support, beloning support, and tangible support). Each dimension is measured by 4 items on a 4-point scale ranging from "Definitely True" to "Definitely False". Total score range 0-36 with a higher score indicating greater social support.
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pulmonary Rehabilitation Program Intervention | Usual Care
Number analyzed (Participants) | 142 | 139
score on a scale | 0.58 [-0.16 to 1.32] | -0.04 [-0.72 to 0.63]
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program Intervention vs Usual Care; Test type: Superiority; p = 0.2216, t-test, 2 sided

7. Secondary Outcome: Meaning in Life
Description: Meaning in Life Questionnaire- 10 item questionnaire measuring the purpose, meaning and presence in life. A higher score indicates a perception of higher meaning and purpose. Scores range from 10-70, a higher score indicates a high perceived meaning and purpose in the respondents life.
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pulmonary Rehabilitation Program Intervention | Usual Care
Number analyzed (Participants) | 144 | 140
score on a scale | 0.07 [-0.68 to 0.82] | -0.33 [-1.13 to 0.48]
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program Intervention vs Usual Care; Test type: Superiority; p = 0.4762, t-test, 2 sided

8. Secondary Outcome: Change in Sleep Quality
Description: Measured using the Pittsburgh Sleep Quality Index to assess severity of sleep disturbances. 9 item questionnaire with total possible scores range from 0 to 21. A lower score suggests a better quality of sleep and a higher score indicates a worse outcome/more severe symptoms of disturbance.
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pulmonary Rehabilitation Program Intervention | Usual Care
Number analyzed (Participants) | 100 | 114
score on a scale | -0.72 [-1.09 to -0.34] | 0.03 [-0.36 to 0.42]
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program Intervention vs Usual Care; Test type: Superiority; p = 0.0068, t-test, 2 sided

9. Secondary Outcome: Change in Anxiety
Description: Measured using the General Anxiety Disorder-2 item Questionnaire screening for anxiety. Score ranges from 0 to 6.,A higher score suggests that anxiety is present.
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pulmonary Rehabilitation Program Intervention | Usual Care
Number analyzed (Participants) | 144 | 142
score on a scale | -0.42 [-0.68 to -0.15] | -0.24 [-0.57 to 0.09]
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program Intervention vs Usual Care; Test type: Superiority; p = 0.1548, t-test, 2 sided

10. Secondary Outcome: Healthcare Utilization
Description: Number of subjects to have an emergency room visits or hospitalization.
Time Frame: 3 months
Population: 46 in the intervention arm were not included in the analysis, 27 withdrew consent, 18 did not complete measures at 3-month and 1 did not complete baseline measures. 45 in the usual care arm were not included in the analysis, 26 withdrew consent, 5 died, and 14 did not complete 3-month measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Pulmonary Rehabilitation Program Intervention | Usual Care
Number analyzed (Participants) | 142 | 142
Participants
  Any Emergency Room Visit | 13 | 24
  Any Hospitalization | 15 | 15

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 9 months on all participants.
Description: This study tracked emergency room and hospitalizations for all causes. None of the ER visits or hospitalizations or deaths were related to this study.
Arm/Group | Pulmonary Rehabilitation Program Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/188 | 5/187
Serious Adverse Events (participants affected / at risk) | 15/188 | 15/187
Other Adverse Events (participants affected / at risk) | 0/188 | 0/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulmonary Rehabilitation Program Intervention (N=188) | Usual Care (N=187)
Hospitalization- COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 9 (14) | 10 (16)
Hospitalization: Aortic Stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization: Opioid Hyperalgesia (General disorders) | 1 (1) | 0 (0)
Hospitalization- left Carotid Artery Stent (Vascular disorders) | 1 (1) | 0 (0)
Hospitalization: Debridement of Metatarsal ulcer (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalization: Endobronchial valve lung volume reduction sugery (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalization: Obstruction Intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hospitalization: Prostate Cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hospitalization: Neoplasm of Rectum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hospitalization: Malignant Neoplasm Brain (Nervous system disorders) | 0 (0) | 1 (1)
Hospitalization: Acute Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hospitalization: Pacemaker Cardiac Status Post (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT03480386/Prot_SAP_000.pdf